CLINICAL TRIAL: NCT01736735
Title: A Phase 2b, Randomized, Double-Blind, Multi-center Study Comparing Cross-linked Polyelectrolyte (CLP) With Placebo in Heart Failure Subjects
Brief Title: Evaluation of Cross-Linked Polyelectrolyte (CLP) With Placebo in Heart Failure Subjects
Acronym: STEPWISE
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sorbent Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CTST-24
Record Dates: First submitted 2012-11-26; First posted 2012-11-29 (Estimated); Last update posted 2014-03-05 (Estimated); Status verified 2014-03

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CLP (Experimental): CLP BID
  Interventions: Drug: CLP
- Placebo (Placebo Comparator): BID powder
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: CLP
  Arms: CLP
Drug: placebo
  Arms: Placebo

SUMMARY:
This is a placebo-controlled study to determine the effect of CLP in heart failure subjects with fluid overload.

ELIGIBILITY:
Selected Inclusion Criteria:

* Age 21 years or older at randomization
* Heart failure with at least one of the following signs of current fluid overload:

  1. Peripheral (or sacral) edema >1+ or ascites during screening or on day of randomization
  2. Pulmonary congestion as determined by chest X-ray during the screening period
* Ambulatory and able to perform the 6-minute walk test

Selected Exclusion Criteria:

* Participation in another clinical trial of an investigational or marketed drug within 30 days or 5 half-lives (whichever is longer) preceding screening
* Any hospitalization or unscheduled outpatient decongestion therapy using IV diuretics, ultrafiltration, or paracentesis within 8 weeks prior to or during screening
* Coronary-artery bypass graft, percutaneous intervention (e.g., cardiac, cerebrovascular, aortic), or major surgery including thoracic and cardiac, within 2 months prior to or during screening or anticipated need during study participation
* Heart transplant recipient, or anticipated need for transplant or LVAD during study participation
* Any of the following events having occurred within 8 weeks prior to or during screening: myocardial infarction, transient ischemic attack, stroke, or acute coronary syndrome as judged by the Investigator

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2013-01; Primary Completion 2014-06 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Composite endpoint comprised of: 6-Minute Walk Test, Body weight, KCCQ Score, Log2 NT-proBNP, time to first occurrence of heart/renal failure hospitalization, unscheduled outpatient intravenous or mechanical therapy for heart/renal failure or death | Baseline, Week 8
  Composite endpoint for the change from baseline to 8 weeks comprised of the following: 6-Minute Walk Test (6 MWT), Body weight, KCCQ Score, Log2 NT-proBNP, time to first occurrence of heart failure or renal failure hospitalization, unscheduled outpatient intravenous or mechanical therapy for heart failure or renal failure, or death.

SECONDARY OUTCOMES:
Change in 6-Minute Walk Test distance from baseline to Week 8. | Baseline, Week 8
Time to heart failure or renal failure hospitalization, unscheduled outpatient intravenous or mechanical therapy for heart failure or renal failure, or death | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Howard Dittrich, MD, Study Chair — Sorbent Therapeutics, Study Sponsor
Locations (3):
- Orange Country Research Center, Tustin, California, United States
- Buenos Aires, Argentina
- Ashkelon, Israel